CLINICAL TRIAL: NCT05406934
Title: Evaluation of Blood Platelet Indices, Platelet Aggregation and Coagulation Profile in the Activity State of Inflammatory Bowel Disease Patients on Biological Treatment
Brief Title: Evaluation of Blood Platelet Indices,Platelet Aggregation in the Activity of IBD Patients on Biological Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maria Hamdy AbdelElmalak, principal investigator, Assiut University
Other Study IDs: AssuitU22
Record Dates: First submitted 2022-01-17; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Bowel Disease; Inflammatory Bowel Diseases
MeSH Terms: conditions — Intestinal Diseases; Inflammatory Bowel Diseases | interventions — Infliximab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- healthy group: the healthy group, not diagnosed IBD
  Interventions: Biological: Infliximab
- IBD patients controlled by conventional treatment: controlled by conventional treatment and divided to UC group and Crohns group
  Interventions: Biological: Infliximab
- uncontrolled IBD patients on biological's treatment: divided to uc received biological and Crohns received biolgical
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — obseravation with investigation

SUMMARY:
ulcerative colitis and Crohn's disease, the two major forms of inflammatory bowel disease, are chronic, idiopathic, relapsing inflammatory conditions of the gastrointestinal tract. The mechanism is multifactorial and may result from the combined interaction of environmental, genetic, epithelial barrier defects, dysregulated immune responses, and microbial factors

DETAILED DESCRIPTION:
Histopathological examinations play a role in the diagnosis and management of UC, but they are costly and invasive. So, non-invasive inflammatory biomarkers of IBD, such as the WBCS, ESR and CRP are used in clinical practice .

Platelets play a critical role in blood hemostasis so impaired platelet activation may cause persistent mucosal inflammation. Many studies have demonstrated that patients with IBD may have increased risks of venous thrombosis. Thrombosis is a major cause of morbidity and mortality in IBD.

Platelet to lymphocyte ratio can be easily calculated from CBC can serve as useful biomarkers for predicting mucosal inflammation in UC.

Current disease management guidelines were focused on the use of anti-inflammatory agents, aminosalicylates, and corticosteroids. However, some patients are still refractory to these therapies.

Biological therapy has revolutionized the management of inflammatory bowel disease in the last few years. There available biologic medicines are infliximab, adalimumab, golimumab, vedolizumab, and ustekinumab. Biological therapy brought a better control of inflammatory bowel diseases. Its use requires specific care before the beginning and during the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. All patients diagnosed with inflammatory bowel disease ulcerative colitis or crohn's disease
2. All IBD patients received biological treatment
3. All IBD patients controlled with conventional treatment

Exclusion Criteria:

1. IBS patients
2. IBD Patients with: a) another autoimmune disease like ITP and SLE B) Bleeding tendency as hemophilia or thrombophilia C) Previous thrombotic events or on anticoagulants or antiplatelet drugs D) With another comorbidity as liver cell failure, respiratory failure, renal failure and cardiac failure

Ages: 21 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: study will include 120 persons divided to 30 healthy persons and 90 was diagnosed inflammatory bowel disease in Asyut university hospital , 60 of those patients diagnosed ulcerative colitis , 30 of them controlled on conventional treatment , 30 patients on biological treatment and 30 patients' crohn's disease , 15 of them controlled on conventional treatment and 15 patients on biological treatment
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-05 (Estimated); Primary Completion 2022-06-05 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
detect of disease activity of IBD patients received biological treatment in the start and in 14 weeks after treatment compared to whose controlled by platelet indices and platelet lymphocytic ratio. | about 14 weeks after start of treatment of inflixmab
  Evaluation of disease activity of IBD patients received biological treatment in the start and in 14 weeks after treatment compared to whose controlled by platelet indices and platelet lymphocytic ratio.

IPD SHARING:
Plan to Share IPD: Undecided